CLINICAL TRIAL: NCT06224790
Title: Effectiveness & Safety of Perfenidone in Type 2 Diabetic Patients With Diabetic Neuropathy: A Randomized Controlled Trial
Brief Title: Perfenidone in Type 2 Diabetic Patients With Diabetic Neuropathy
Acronym: PenDaNt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sidrah Lodhi (Other)
Responsible Party: Sponsor-Investigator, Sidrah Lodhi, Assistant Professor of Medicine, King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 483/RC/KEMU/2022
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Nephropathies; Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Perfenidone
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Pirfenidone) (Experimental): Capsule Pirfenidone 200mg, 2 X 8hrly for 3 months
  Interventions: Drug: Pirfenidone
- Group B (Placebo Comparator): Placebo capsules - 2 X 8hrly for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Capsule Pirfenidone 1200mg/ day in divided doses for 3 months
  Arms: Group A (Pirfenidone)
Other: Placebo — 2 Capsules 3 times a day for 3 months
  Arms: Group B

SUMMARY:
The purpose of this study is to determine the effectiveness & safety of pirfenidone in type 2 diabetic patients with diabetic nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Nephropathy Stage 3 (eGFR 30-59 mL/min/1.73m2) Type 2 Diabetes HbA1c <7.5% Patient taking ACEi/ARB for at least 3 months BP <140/90

Exclusion Criteria:

* History of photosensitivity rash History of decompensated liver or cardiac disease History of urinary tract infection Pregnancy or lactation History of nephrotoxic drugs or hakeem medication Polycystic kidney disease History of autoimmune disease History of hypersensitivity to study drugs

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
15% improvement in eGFR | 6 months
  eGFR of the patients shall be evaluated for at least 15% improvement

SECONDARY OUTCOMES:
Safety - Adverse Effects of Drugs | 6 months
  Adverse Effects of the drugs

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No